CLINICAL TRIAL: NCT04426383
Title: Evaluation of a TDM Program for Intensive Care Patients in the Cerebrospinal
Brief Title: Evaluation of a TDM Program for Intensive Care Patients in the Cerebrospinal Fluid
Acronym: EMIL
Status: Completed | Type: Observational
Sponsor: Ludwig-Maximilians - University of Munich (Other)
Collaborators: Freie Universität Berlin (Other)
Responsible Party: Principal Investigator, Michael Zoller MD, senior physician, Department of Anaesthesiology, university hospital munich, Ludwig-Maximilians - University of Munich
Other Study IDs: LMU 20-169
Record Dates: First submitted 2020-06-04; First posted 2020-06-11 (Actual); Last update posted 2022-06-01 (Actual); Status verified 2022-05

CONDITIONS: Ventriculitis, Infectious
Keywords: therapeutic drug monitoring (TDM); critically ill patients; cerebrospinal fluid
MeSH Terms: conditions — Cerebral Ventriculitis

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 28 Days
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
Therapeutic drug monitoring of antibiotics in critically ill patients is a present research topic of the last ten years. Research results have shown subtherapeutic blood concentrations in those patients. However, the amount of antibiotics in the cerebrospinal fluid (CSF) in patients with ventriculitis or meningitis is still unclear. This study is a prospective study to evaluate the concentration of different antibiotics in the CSF in patients with an external ventricular drainage compared to antibiotic blood concentration.

DETAILED DESCRIPTION:
Bacterial infections are still associated with a high mortality in intensive care unit patients. Especially patients diagnosed with ventriculitis caused by a bacterial infection have a bad outcome. Therefore, antibiotic therapy is the only causal opportunity to treat those infections. However, there are many chances in pharmacokinetic and -dynamic in critically ill patients with unpredictable antibiotic concentrations. Furthermore, it is important that the concentration in the blood as well as in the effect-compartment "CSF" is sufficient. Less data of the last years describe antibiotic concentrations in the CSF and show subtherapeutic levels, which is endangering for the therapeutic success. The introduced study is a prospective, observational study that analyses antibiotic concentrations in CSF in critically ill patients. The distribution between CSF and blood will be evaluated by comparing these two compartments.

ELIGIBILITY:
Inclusion Criteria:

* written approval of the legal guardian
* external ventricular drainage
* antibiotic therapy

Exclusion Criteria:

* no approval
* no antibiotic therapy or no external ventricular drainage

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: critically ill patients with an external ventricular drainage and the need of antibiotic therapy
Sampling Method: Probability Sample
Enrollment: 32 (Actual)
Dates: Start 2020-06-01 (Actual); Primary Completion 2022-01-31 (Actual); Study Completion 2022-05-01 (Actual)

PRIMARY OUTCOMES:
Incidence of subtherapeutic antibiotic concentrations in cerebrospinal fluid | through study completion, on average 2 years
  Percentage of subtherapeutic concentrations of different antibiotics in different subgroups like ventriculitis vs. no ventriculitis

SECONDARY OUTCOMES:
28-day mortality | through study completion, on average 2 years
  evaluation of the 28-day mortality in patients with therapeutic and subtherapeutic antibiotic concentrations in cerebrospinal fluid
Correlation of antibiotic concentration in cerebrospinal fluid and C-reactive protein | through study completion, on average 2 years
  Correlation of different antibiotic concentrations in patients´ blood and cerebrospinal fluid and the C-reactive protein in the blood. Question of interest is, if therapeutic antibiotic concentration leads to a faster decrease of C-reactive protein
Correlation of antibiotic concentration in cerebrospinal fluid and interleucin 6 | through study completion, on average 2 years
  Correlation of different antibiotic concentrations in patients´ blood and cerebrospinal fluid and the interleucin 6 in the blood. Question of interest is, if therapeutic antibiotic concentration leads to a faster decrease of interleucin 6

CONTACTS AND LOCATIONS:
Overall Officials: Michael Zoller, Principal Investigator — Ludwig-Maximilians - University of Munich
Locations (1):
- Department of Anaesthesiology of the University Hospital of Munich, Munich, Germany

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Wicha SG, Kinast C, Munchow M, Wittova S, Greppmair S, Kunzelmann AK, Zoller M, Paal M, Vogeser M, Habler K, Weig T, Terpolilli N, Heck S, Dimitriadis K, Scharf C, Liebchen U. Meropenem pharmacokinetics in cerebrospinal fluid: comparing intermittent and continuous infusion strategies in critically ill patients-a prospective cohort study. Antimicrob Agents Chemother. 2024 Sep 4;68(9):e0045124. doi: 10.1128/aac.00451-24. Epub 2024 Jul 31. PMID 39082803
- [Derived] Chen Z, Taubert M, Chen C, Dokos C, Fuhr U, Weig T, Zoller M, Heck S, Dimitriadis K, Terpolilli N, Kinast C, Scharf C, Lier C, Dorn C, Liebchen U. Plasma and Cerebrospinal Fluid Population Pharmacokinetics of Vancomycin in Patients with External Ventricular Drain. Antimicrob Agents Chemother. 2023 Jun 15;67(6):e0024123. doi: 10.1128/aac.00241-23. Epub 2023 May 10. PMID 37162349